CLINICAL TRIAL: NCT07166835
Title: The Efficacy of a Blackcurrant-based Nootropic Drink to Support Cognitive Functioning Under Normobaric Simulated High Altitude
Brief Title: Exploring the Cognitive Benefits of a Blackcurrant-Based Supplement in Normobaric Hypoxia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Leeds Beckett University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 151421
Record Dates: First submitted 2025-08-26; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Cognitive Performance; Executive Function (Cognition); Working Memory; Hypoxia Induced Cognitive Impairment; Mood
MeSH Terms: interventions — Nootropic Agents; Ginkgo Extract; Nicergoline; Piracetam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nootropic drink (Active Comparator): Nootropic beverage containing anthocyanins, L-theanine, and Enzogenol. Administered orally prior to cognitive testing under simulated normobaric hypoxia.
  Interventions: Dietary Supplement: Nootropics (ginkgo biloba, nicergoline, piracetam, or others)
- Placebo drink (Placebo Comparator): Taste- and appearance-matched placebo beverage without active ingredients. Administered orally prior to cognitive testing under simulated normobaric hypoxia.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Nootropics (ginkgo biloba, nicergoline, piracetam, or others) — Nootropic drink containing Anthrocyanins, L-theanie and Enzogenol
  Arms: Nootropic drink
Dietary Supplement: Placebo — Taste- and appearance-matched placebo beverage without active ingredients.
  Arms: Placebo drink

SUMMARY:
This study investigates the cognitive effects of Ārepa, a blackcurrant-based drink, under simulated high-altitude conditions (4,500m normobaric hypoxia for ~180 minutes). Using a double-blind, randomised, placebo-controlled crossover design, participants will consume either the nootropic blackcurrant-based drink or a taste-matched placebo. Cognitive testing (~80 minutes) includes Trail-making, Stroop, N-back, Serial 7s/3s, and RVIP tasks. Physiological measures (heart rate, SpO₂, blood) and biomarkers (MAO-B, BDNF, hsCRP, S100B, Prolactin, C3G, Sarmentosin) will be assessed. Scales will evaluate mood, wellbeing, and perceived effects. The aim is to determine if the nootropic drink can support cognitive function in hypoxic environments.

DETAILED DESCRIPTION:
Cognitive functioning can be influenced by varying factors including age, education, fatigue and environmental conditions. It is well established that stress, including hypoxia, sleep deprivation, and mental fatigue, alters brain energetics therefore resulting in a decline of cognitive function. Any physical or psychological stressor that disrupts homeostasis results in a stress response. Altitude, often associated with sports, recreational activities and holidaying, refers to environments where the partial pressure of oxygen (pO2) is reduced relative to sea level. The effects of high altitude on humans are mostly the consequences of reduced pO2 in the atmosphere and can result in fatigue, dizziness and debilitating cognitive consequences to unacclimatised individuals. These effects can significantly impair cognitive and physical performance at high elevations. In this context, interests in prophylactic use of dietary interventions to mitigate the effects of oxygen deprivation has increased in recent years. Interventions utilising a number of plant derived phytochemicals have demonstrated some protective efficacy against these physiological insults and may be capable of attenuating cognitive function and mood under hypoxic stress. However, there is limited research available on polyphenol supplementation to support cognition at high altitudes. Therefore, the purpose of the study is to explore the possibility of the nootropic drink and how effective it is in reducing cognitive impairment of healthy males at a simulated high altitude of 4,500m.

Participants will attend the laboratory on four occasions over a 2-3-week period. The first two visits will involve a pre-screening assessment and a familiarisation session with the experimental procedures and cognitive tasks.

The subsequent two visits will serve as the experimental trials, during which participants will be exposed to a normobaric hypoxic environment simulating an altitude of 4,500 meters. This condition is achieved by maintaining sea-level barometric pressure with a reduced inspired oxygen fraction (FiO₂ ~11.3%, equivalent to a PiO₂ of approximately 80.9 mmHg).

Acute exposure to high altitudes (3,000-4,500 m) for durations as short as 45 to 120 minutes has been shown to impair cognitive function, increase mood disturbances, reduce task accuracy, and slow reaction times. Based on prior research the duration of hypoxic exposure in this study will be approximately 180 minutes, allowing sufficient time for potential cognitive changes to occur.

Each experimental trial will follow a double-blind, randomised, placebo-controlled crossover design. Participants will consume 100 mL of either an anthocyanin-rich blackcurrant drink (containing 200 mg of bioactive compounds) or a taste- and appearance-matched placebo (0 mg). A 45-minute rest period will follow to allow for absorption.

Cognitive testing will span approximately 80 minutes and will begin 75 minutes into the hypoxic exposure. This includes three short tasks (approximately 10 minutes in total) administered before and after a 60-minute cognitive demand battery. The cognitive tasks will assess executive function, working memory, attention, and cognitive load.

Physiological measures (e.g., heart rate, SpO₂), blood-based biomarkers (e.g., MAO-B, BDNF, hsCRP, S100B, prolactin, C3G, sarmentosin), and self-reported scales assessing mood, anxiety, perceived cognitive workload, and subjective effects will also be collected throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent (in English)
* Aged 18-35
* Male
* Residing at a low altitude (<500m)

Exclusion Criteria:

* Diagnosed food allergy or intolerance to the investigational products or control products. (Blackcurrant, food allergen/ pine, tree-derived allergen/ l-theanine tree allergen (camellia sinensis))
* Significant past medical and psychiatric history and ongoing chronic conditions such as, cardiovascular disease, respiratory disease, endocrine disorder (e.g. Diabetes mellites) and neurological and psychiatric conditions including brain injury or are colourblind.
* Significant medication history or current prescription of medication or supplements known to affect cognition such as. Sedatives, stimulants, or herbal supplements high in anthocyanin and polyphenol content.
* A positive result from the pre-screening sickle cell trait blood test.
* An abnormal ECG reading.
* A resting heart rate above 100bmp.
* A blood pressure reading above 140/90mmHg.
* Subjects not willing and/ or not able to comply with the scheduled visits required for the study.
* Not willing to provide blood samples.
* Not classified as low risk based on the ACSM guidelines.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — cisgendered men
Enrollment: 27 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-12-25 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Executive Function (Trail Making Task) | Baseline (sea level, pre-supplementation), approximately 1 hour (±10 minutes) after exposure, and 2 hours (±10 minutes) after exposure.
  Change from baseline (sea level, pre-supplementation) in completion time during acute high-altitude exposure, assessed at ~1 hour and ~2 hours post exposure following a cognitive demand battery. Measures of correct response and reaction time in seconds.
Working Memory (N-back) | Baseline (sea level, pre-supplementation), approximately 1 hour (±10 minutes) after exposure, and 2 hours (±10 minutes) after exposure.
  Change from baseline (sea level, pre-supplementation) in accuracy (percent correct responses) and mean reaction time (milliseconds) on the N-back task during acute high-altitude exposure, assessed at ~1 hour and ~2 hours post exposure following a cognitive demand battery. Measures are response time in milliseconds and percentage of correct response.
Attention (RVIP) as part of the Cognitive Demand Battery | Baseline (sea level, pre-supplementation), and 6 repeated assessments during the cognitive demand battery conducted between 1 hr 20 min and 2 hr 20 min after onset of acute high-altitude exposure.
  Change from baseline (sea level, pre-supplementation) in accuracy (percent correct) and mean reaction time (milliseconds) on the RVIP task, administered as part of a repeated cognitive demand battery beginning ~1 hr 20 min into acute high-altitude exposure and repeated 6 times within 1 hour.
Executive Function (Stroop, colour word task) | Baseline (sea level, pre-supplementation), approximately 1 hour (±10 minutes) after exposure, and 2 hours (±10 minutes) after exposure.
  Change from baseline (sea level, pre-supplementation) in number of correct responses and mean reaction time during acute high-altitude exposure, assessed at ~1 hour and ~2 hours post exposure following a cognitive demand battery. Measures are number of correct responses and response time in seconds.
Working Memory (Serial 7s) | Baseline (sea level, pre-supplementation), and 6 repeated assessments during the cognitive demand battery conducted between 1 hr 20 min and 2 hr 20 min after onset of acute high-altitude exposure.
  Change from baseline (sea level, pre-supplementation) in number of correct subtractions on the Serial 7s task, administered as part of a repeated cognitive demand battery beginning ~1 hr 20 min into acute high-altitude exposure and repeated 6 times within 1 hour. Measure is Number of correct responses.
Working Memory (Serial 3s) | Baseline (sea level, pre-supplementation), and 6 repeated assessments during the cognitive demand battery conducted between 1 hr 20 min and 2 hr 20 min after onset of acute high-altitude exposure.
  Change from baseline (sea level, pre-supplementation) in number of correct subtractions on the Serial 3s task, administered as part of a repeated cognitive demand battery beginning ~1 hr 20 min into acute high-altitude exposure and repeated 6 times within 1 hour. Units of measure is the number of correct responses.

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds Beckett University, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No